CLINICAL TRIAL: NCT04062409
Title: Effect of Salbutamol on Autonomic Nervous System Dysfunction of Children With Sickle Cell Disease
Brief Title: Autonomic Nervous System and Sickle Cell Disease
Acronym: DrepaSympa
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K170302
Record Dates: First submitted 2019-08-19; First posted 2019-08-20 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2019-08

CONDITIONS: Heart Rate Variability (ANS Function)
Keywords: sickle cell disease; asthma; beta-agonist; hear rate variability
MeSH Terms: conditions — Anemia, Sickle Cell; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sickle cell patients
- Asmathic patients

SUMMARY:
Sickle cell disease (SCD) children and adults with asthma have an increased rate of vaso-occlusive crisis, acute chest syndrome episodes, and premature mortality when compared to those without asthma. We hypothesised that either asthma diagnosis and/or bronchodilator treatment may aggravate SCD via their modulating effect on autonomic nervous system.

DETAILED DESCRIPTION:
Heart rate variability during pulmonary function tests (spirometry, static volumes, DLCO/DLNO, exhaled NO at multiple flow rates) including salbutamol administration will be evaluated in patients with SCD (n=60) receiving asthma treatment or not, as compared to asthmatic children without SCD (n=30) matched for ethnicity

ELIGIBILITY:
Inclusion Criteria:

* age from 8 to 16 years (≥ 8 years and < 16 years) (spirometry and DLCO study feasible)
* Sub-Saharan African or Caribbean ethnic origin.
* child with sickle cell disease referred for monitoring of respiratory function in the framework of its sickle cell disease and whether or not it presents a possible disease asthmatic (asthma treatment prescribed in the past year)
* or asthmatic child (typical functional signs + history of exacerbation severe hospitalized or reversible obstructive pulmonary disorder) not sickle cell
* addressed for respiratory function monitoring

Exclusion Criteria:

* Refusal to participate (lack of consent)
* Sickle cell child of North African origin

Ages: 6 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Subjects of African or Caribbean ethnicity who were 8 to 16 years of age and were referred to the Pulmonary function Testing unit for the follow-up of their disease : SCD or asthma
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
To assess the effect of salbutamol administration on ANS in these SCD children (with and without asthma) and in control asthmatics (without SCD) | cross-sectional, one hour
  heart rate variability after salbutamol administration

SECONDARY OUTCOMES:
To assess ANS functions in patients with SCD receiving asthma treatment or not, as compared to asthmatic children without SCD matched for ethnicity | cross-sectional, one hour
  baseline heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Delclaux, MD PhD, Principal Investigator — APHP
Locations (1):
- Robert Debre Hospital, Paris, France

REFERENCES:
- [Result] Bokov P, El Jurdi H, Denjoy I, Peiffer C, Medjahdi N, Holvoet L, Benkerrou M, Delclaux C. Salbutamol Worsens the Autonomic Nervous System Dysfunction of Children With Sickle Cell Disease. Front Physiol. 2020 Feb 26;11:31. doi: 10.3389/fphys.2020.00031. eCollection 2020. PMID 32174840